CLINICAL TRIAL: NCT06301295
Title: Feasibility of Targeted Bronchial Washing Fluid for Molecular Testing With Next Generation Sequencing in Patients With Early-stage Non-small Cell Lung Cancer
Brief Title: Feasibility of Targeted Bronchial Washing for Molecular Testing by Next Generation Sequencing in Early-stage Lung Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2402-017-136
Record Dates: First submitted 2024-03-03; First posted 2024-03-08 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer
Keywords: Bronchoscopy; Liquid biopsy; Lung Cancer; Next Generation Sequencing
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrathin bronchoscopy with intratumoral washing (Experimental): Each subject suspected of early-stage lung cancer will undergo bronchooscopic procedure for generic alteration with Next Generation Sequencing.
  Interventions: Diagnostic Test: Ultarthin bronchoscopy with intratumoral washing

INTERVENTIONS:
Diagnostic Test: Ultarthin bronchoscopy with intratumoral washing — Each subject suspected of early-stage, resectable lung cancer will undergo bronchooscopic procedure. Ultrathin bronchoscope is inserted and placed within tumor under radial EBUS, virtual bronchoscopic navigation, and fluoroscopy guidance. Subsequently, intratumoral washing is performed. After undergoing surgery for suspected early-stage lung cancer, the analysis of next generation sequencing is conducted on intratumoral washing, tissue from surgical specimen, and blood.

SUMMARY:
This is a single center, clinical trial evaluating the relevance of intratumoral washing for detection of generic alteration with Next Generation Sequencing.

DETAILED DESCRIPTION:
This is a prospective, single-arm, open-label study to assess evaluate the relevance of intratumoral washing by ultrathin bronchoscopy (outer diameter; 3mm) for detection of genetic alterations using Next Generation Sequencing in patients suspicious of early-stage lung cancer.

ELIGIBILITY:
1. Inclusion Criteria:

   * Age ≥ 20 years
   * Obtained written informed consent
   * Subjects suspected of having resectable lung cancer on computed tomography
   * Subjects without contraindication to brochoscopy
   * Subjects planning to undergo surgery for suspected lung cancer and opting for tissue or liquid biopsy for genetic alteration using Next Generation Sequencing
2. Exclusion Criteria:

   * Subjects who withdraw informed consent
   * Subjects who are unable to undergo liquid biopsy (plasma) and tissue biopsy - for genetic alteration with Next Generation Sequencing based on the investigator's judgement
   * Subjects diagnosed with a cancer other than non-small cell lung cancer from the lung tissue lesion
   * Subjects diagnosed with a benign lesion from the lung tissue lesion

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The diagnostic accuracy of genetic alterations in intratumoral washing fluid using Next Generation Sequencing | through study completion, an average of 1 year
  Diagnostic accuracy is defined as the number of true positive and true negative genetic alterations detected by Next Generation Sequencing, divided by the total number of intratumoral washing attempts using ultrathin bronchoscopy.

SECONDARY OUTCOMES:
Detection rate of clinically significant actionable mutations among intratumoral washing fluid, plasma, and tissue | through study completion, an average of 1 year
  Detection rate is defined as the number of genetic alterations detected by Next Generation Sequencing divided by the total number of intratumoral washing attempts using ultrathin bronchoscopy. Clinically significant actionable mutations are defined as genes with corresponding drugs, either approved or under clinical trial (e.g., EGFR, ALK, ROS1, BRAF V600E, RET, NTRK, KRAS G12C, FGFR3, or HER2).
Concordance rate of genetic alterations detected by Next Generation Sequencing among intratumoral washing fluid, plasma, and tissue | through study completion, an average of 1 year
  The concordance rate of genetic alterations detected by Next Generation Sequencing in intratumoral washing fluid, compared with plasma and tissue (gold standard).
Sensitivity and specificity of genetic alterations detected by Next Generation Sequencing in intratumoral washing fluid | through study completion, an average of 1 year
  The sensitivity and specificity of genetic alterations detected by Next Generation Sequencing in intratumoral washing fluid compared with tissue (gold standard).
Turn-around time | through study completion, an average of 1 year
  The duration between an order request and the task completion in in intratumoral washing fluid compared with plasma and tissue (gold standard).
Detection rate of co-mutations among intratumoral washing fluid, plasma, and tissue | through study completion, an average of 1 year
  Detection rate is defined as the number of genetic alterations detected by Next Generation Sequencing divided by the total number of intratumoral washing attempts using ultrathin bronchoscopy. Co-mutations are defined as the occurrence of two or more genetic alterations within the same tumor cells in an individual, including at least one actionable mutation (e.g., TP53, DNMT3A, TET2, CTNNB1, PIK3CA, RB1, STK11).

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Seop Eom, MD, PhD, Principal Investigator — Pusan National University Hospital
Locations (1):
- Pusan National University Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No